CLINICAL TRIAL: NCT02282163
Title: A Multicenter Clinical Evaluation of Safety and Efficacy of Lumason as a Contrast Agent in Pediatric Echocardiography
Brief Title: Evaluation of Safety and Efficacy of Lumason in Pediatric Echocardiography
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA agreed to early termination due to difficulties enrolling patients.
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BR1-140
Record Dates: First submitted 2014-10-30; First posted 2014-11-04 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases | interventions — contrast agent BR1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lumason (Experimental): All patients were administered, Lumason (sulphur hexafluoride lipid-type A microspheres) an ultrasound contrast agent as a single 0.03 mL/kg bolus injection during echocardiography.
  Interventions: Drug: sulphur hexafluoride lipid-type A microspheres

INTERVENTIONS:
Drug: sulphur hexafluoride lipid-type A microspheres — Ultrasound imaging contrast agent
  Other Names: Lumason; SonoVue

SUMMARY:
Safety and Efficacy Study in pediatric subjects aged 9 to 17 years of age with suboptimal LV EBD on non-contrast 2D echocardiography. Imaging modalities that are used throughout the study in pediatric subjects represented those utilized in routine clinical practice in adults.

DETAILED DESCRIPTION:
This was a Phase III, multicenter, open-label study that was to be conducted at approximately 7-12 sites in the United States, Canada and Europe in pediatric patients with suboptimal LV EBD on non-contrast 2D transthoracic echocardiography. It was estimated that 92 patients were to be enrolled to provide 73 evaluable patients.

Three cardiologists unaffiliated with enrolling centers (blinded readers), blinded to the patient's identity and clinical profile were to independently evaluate the echocardiograms. The efficacy analysis was primarily based on the blinded reader evaluations.

Imaging modalities that are used throughout the study in pediatric subjects represented those utilized in routine clinical practice in adults.

One of the sites participating in this study was to be asked to consent a subset of patients for additional blood sampling for analysis of SF6 concentration in blood from a total of 6 patients (3 males and 3 females) in the age group 9 up to 12 years of age and 6 patients (3 males and 3 females) in the age of >12 up to and including 17 years.

The current study was designed to assess the efficacy of Lumason-enhanced echocardiography in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Provide Written informed consent from parent(s) or legal guardian
* Provide assent when required according to local regulations
* Suspected of having cardiac disease or undergoing evaluation of cardiac anatomy for congenital heart disease
* Undergone a previous transthoracic echocardiogram within one month prior to enrollment resulting in suboptimal left ventricular endocardial border defined as ≥ 2 contiguous segments in any given view that cannot be visualized.

Exclusion Criteria:

* Children < 9 years of age
* Previously enrolled in the study
* Administered any other contrast agent either intravascularly or orally within 48 hours of Lumason administration
* Known right-to-left, bidirectional or transient cardiac shunt (ruled out with agitated saline study performed before administration of Lumason)
* Known hypersensitivity to one or more of the ingredients of the investigational product
* Received an investigational compound within 30 days before enrolling into this study
* Pregnant or lactating female
* Determined by investigator to be unsuitable for the study

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melda Dolan, M.D., Study Director — Bracco Diagnostics, Inc
Locations (2):
- United States (2):
  - Washington University School of Medicine in Saint Louis, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Initiation Date (first subject enrolled): 20 October 2015; Study Completion Date (last subject completed study related activities): 20 January 2018. Enrolment was at 2 sites in the US.
  Even though last subject enrolled was 20 January 2018, FDA release from completion of enrolment was 31 May 2018. Blinded read completion was 13 August 2018.
Pre-assignment Details: The study was terminated early due to challenges with enrollment. At the time of termination, 13 subjects were enrolled and 12 subjects were dosed with Lumason, thus the efficacy analysis was considered as exploratory and p-values are not included in the Results section.
  PK assessment was not performed due to enrollment difficulties.
Period: Overall Study
Arm/Group | Lumason
Started | 13
Completed | 12
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lumason
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (2.29)
Age, Customized [Count of Participants; unit: Participants]
  Age group: 6 to 9 years | 1
  Age group: 10 to 11 years | 0
  Age group: 12 to 15 years | 8
  Age group: 16-17 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 10
  Black | 2
  Asian | 0
  Other | 0
Height [Mean (Standard Deviation); unit: cm] | 156.1 (28.51)
Weight [Mean (Standard Deviation); unit: kg] | 60.76 (23.846)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.35 (12.092)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Left Ventricular Endocardial Border Delineation (LV EBD) Scores
Description: The total LV EBD score for a subject was the total of the EBD scores (Inadequate - 0, sufficient - 1, Good - 2) from the 17 segments (from the apical 4-chamber, apical 2-chamber and apical long (3-chamber) views, according to the guidelines of the American Society of Echocardiography). The total LV EBD scores could range from 0 to 34 and are presented below for each of the three readers for both unenhanced ultrasound (UEUS) and contrast-enhanced ultrasound (CEUS).
  Change from baseline is the difference between UEUS and CEUS in total LV EBD scores.
Time Frame: Immediately post dose-Day 1
Population: All subjects who received IP and had data available for both unenhanced ultrasound (UEUS) and contrast-enhanced ultrasound (CEUS) were included in ITD population.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Off-site Reader 1 UEUS: Off-site Reader 1 UEUS Assessment
- Off-site Reader 1 CEUS: Off-site Reader 1 CEUS Assessment
- Off-site Reader 2 UEUS: Off-site Reader 2 UEUS Assessment
- Off-site Reader 2 CEUS: Off-site Reader 2 CEUS Assessment
- Off-site Reader 3 UEUS: Off-site Reader 3 UEUS Assessment
- Off-site Reader 3 CEUS: Off-site Reader 3 CEUS Assessment
Arm/Group | Off-site Reader 1 UEUS | Off-site Reader 1 CEUS | Off-site Reader 2 UEUS | Off-site Reader 2 CEUS | Off-site Reader 3 UEUS | Off-site Reader 3 CEUS
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12
score on a scale | 6.4 [2.9 to 10.0] | 33.5 [32.6 to 34.3] | 10.6 [6.8 to 14.4] | 33.3 [31.8 to 34.9] | 7.3 [4.0 to 10.5] | 33.0 [31.8 to 34.2]

2. Primary Outcome: Percentage of Participants With Adequate Left Ventricular Opacification (LVO)
Description: LVO was graded as 0 to +3, 4-point rating scale. Left ventricular opacification rating of +2 (non-homogeneous) or +3 (complete and homogeneous) was considered as adequate LVO.
Time Frame: Immediately post dose-Day 1
Population: All subjects who received IP and had data available for contrast-enhanced ultrasound (CEUS) were included in ITD population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Off-site Reader 1 CEUS: Off-site Reader 1 CEUS
- Off-site Reader 2 CEUS: Off-site Reader 2 CEUS
- Off-site Reader 3 CEUS: Off-site Reader 3 CEUS
Arm/Group | Off-site Reader 1 CEUS | Off-site Reader 2 CEUS | Off-site Reader 3 CEUS
Number analyzed (Participants) | 12 | 12 | 12
percentage of participants | 100 [73.5 to 100] | 100 [73.5 to 100] | 100 [73.5 to 100]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: To obtain safety data in pediatric subjects administered Lumason for LV EBD improvement during echocardiography
Time Frame: Up to 72 hours post dose
Population: Summary of adverse events in the safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Lumason
Number analyzed (Participants) | 12
Participants
  Number of Subjects With at Least 1 AE | 5
  Number of Subjects With AEs by Intensity - Mild | 4
  Number of Subjects With AEs by Intensity -Moderate | 1
  Number of Subjects With AEs by Intensity -Severe | 0

ADVERSE EVENTS:
Time Frame: Subjects were monitored for any untoward medical events from the time of signed Informed Consent through 72 hours after IP administration.
Arm/Group | Lumason
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumason (N=12)
Vomiting (Gastrointestinal disorders) | 1 (1)
Injection site bruising (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Abnormal behavior (Psychiatric disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT02282163/Prot_SAP_000.pdf